CLINICAL TRIAL: NCT04839198
Title: Using Machine Learning to Develop Just-in-Time Adaptive Interventions for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Emily Hebert, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-20-1159; R00DA046564 (NIH)
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-09

CONDITIONS: Smoking Cessation
Keywords: Nicotine patch
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adaptive Treatment plus usual care (Experimental)
  Interventions: Behavioral: Android Wear smartwatch; Behavioral: Adaptive Treatment; Drug: Nicotine Patch; Behavioral: interviewing-based counseling
- Usual care (Active Comparator)
  Interventions: Behavioral: Android Wear smartwatch; Drug: Nicotine Patch; Behavioral: interviewing-based counseling

INTERVENTIONS:
Behavioral: Android Wear smartwatch — All participants will wear an Android Wear smartwatch, and will complete ecological momentary assessments (EMA).
Behavioral: Adaptive Treatment — Participants will have access to a "Dashboard" button in the InsightTM app that displays personalized statistics based on their progress and patterns in the study.The dashboard will update as more data is collected about the participant's smoking habits, starting in the pre-quit period and continuing through the post-quit period. Second, in the post-quit period, participants will receive treatment messages when the machine learning algorithm determines that they are at high risk for lapse.At the follow-up visit, participants will complete a survey to evaluate what they liked and disliked about the intervention, how accurate they thought the app was in predicting their risk, and how useful they found the dashboard.
  Arms: Adaptive Treatment plus usual care
Drug: Nicotine Patch — At Visit 2, participants will be asked to begin their attempt to quit smoking and will receive a 12-week supply of nicotine replacement therapy (i.e., nicotine patches and gum)
Behavioral: interviewing-based counseling — At Visit 2, participants will be asked to begin their attempt to quit smoking and meet with a Tobacco Treatment Specialist, who will provide motivational interviewing-based counseling, help the participants develop a quit plan, and discuss relapse prevention. During the 6-weeks of the study, participants will have the option of attending up to 6 counseling sessions with the Tobacco Treatment Specialist, either in-person or via phone or web.

SUMMARY:
The purpose of this study is to evaluate the feasibility and preliminary effectiveness of delivering a personalized, just-in-time adaptive intervention driven by machine learning prediction of smoking lapse risk in real time.

ELIGIBILITY:
Inclusion Criteria:

* a score greater than or equal to 4 on the Rapid Estimate of Adult Literacy in Medicine Short Form (REALM-SF),12
* willingness to quit smoking 14 days after the baseline visit
* no contraindications to using Nicotine replacement therapy (NRT).
* If participants would like to use their own phone to complete the EMAs, they must additionally have an Android smartphone (Android 5.2 or higher), and be willing to install the InsightTM mHealth app on their phone.

Exclusion Criteria:

* currently smoking less than 5 cigarettes per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Number of patients who quit smoking as confirmed by absence of salivary cotinine | 4-weeks after quit day

CONTACTS AND LOCATIONS:
Overall Officials: Emily Hebert, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No